CLINICAL TRIAL: NCT04477512
Title: A Phase 1b Clinical Trial of Cabozantinib and Abiraterone With Checkpoint Inhibitor Immunotherapy in Metastatic Hormone Sensitive Prostate Cancer (CABIOS Trial)
Brief Title: Cabozantinib and Abiraterone With Checkpoint Inhibitor Immunotherapy in Metastatic Hormone Sensitive Prostate Cancer (CABIOS Trial)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202009082
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Hormone Refractory Prostate Cancer
MeSH Terms: interventions — cabozantinib; Nivolumab; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Level 1: Cabozantinib+Abiraterone acetate +Nivolumab (Experimental): -Abiraterone acetate is an oral medication given at a dose of 1000 mg daily. Prednisone is an oral medication given at a dose of 5 mg daily. Nivolumab is given intravenously over 30 minutes on Day 1 of each 28-day cycle at a dose of 480 mg. Cabozantinib is an oral drug given daily; dosing will be 20 mg. Participants can continue to receive treatment for up to 2 years.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Abiraterone acetate; Drug: Prednisone; Procedure: Peripheral blood collection
- Level 2: Cabozantinib+Abiraterone acetate +Nivolumab (Experimental): -Abiraterone acetate is an oral medication given at a dose of 1000 mg daily. Prednisone is an oral medication given at a dose of 5 mg daily. Nivolumab is given intravenously over 30 minutes on Day 1 of each 28-day cycle at a dose of 480 mg. Cabozantinib is an oral drug given daily; dosing will be 40 mg. Participants can continue to receive treatment for up to 2 years.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Abiraterone acetate; Drug: Prednisone; Procedure: Peripheral blood collection
- Expansion: Cabozantinib+Abiraterone acetate +Nivolumab (Experimental): -Abiraterone acetate is an oral medication given at a dose of 1000 mg daily. Prednisone is an oral medication given at a dose of 5 mg daily. Nivolumab is given intravenously over 30 minutes on Day 1 of each 28-day cycle at a dose of 480 mg. Cabozantinib is an oral drug given daily; dosing will be dependent on recommended dose found in first part of study. Participants can continue to receive treatment for up to 2 years.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Abiraterone acetate; Drug: Prednisone; Procedure: Peripheral blood collection

INTERVENTIONS:
Drug: Cabozantinib — Supplied by Exelixis
Drug: Nivolumab — Supplied by Bristol-Myers Squibb
Drug: Abiraterone acetate — Commercially available
Drug: Prednisone — Commercially available
Procedure: Peripheral blood collection — Prior to start of treatment, after 8 weeks of combination therapy, with every subsequent imaging (every 12 weeks), end of treatment

SUMMARY:
The goal of this study is to determine the recommended phase 2 dose of the multi-drug combination of abiraterone, cabozantinib, and nivolumab in conjunction with ongoing androgen deprivation therapy in previously untreated metastatic hormone-sensitive prostate cancer patients. The investigators hypothesize that the combination of cabozantinib and abiraterone acetate/prednisone in conjunction with nivolumab will have an acceptable safety profile and will be feasible to administer in patients with hormone-sensitive metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hormone-sensitive prostate adenocarcinoma.
* Must have evidence of metastatic disease on CT or MRI of the chest, abdomen, and pelvis, or technetium bone scan. May have any type or location of metastases (bone, lymph node, visceral). May have relapsed metastatic disease after initial primary therapy or de novo metastatic disease. Metastatic disease does not have to be confirmed by biopsy.
* May have been on androgen deprivation therapy (ADT) for metastatic hormone-sensitive prostate cancer for ≤ 12 weeks prior to study enrollment (GnRHR agonist such as leuprolide, goserelin, triptorelin, buserelin, histrelin; GnRHR antagonists such as degarelix, or relugolix). Prior ADT for localized prostate cancer is allowed.
* Prior palliative radiation therapy for bone metastasis (must be complete ≥14 days prior to enrollment) or any other radiation therapy (must be complete ≥28 days prior to enrollment) is allowed. Prior definitive radiation therapy for localized prostate cancer is allowed.
* If the patient has undergone bilateral orchiectomy, it must have occurred no more than 12 weeks before study enrollment.
* Recovery to baseline or ≤ grade 1 from toxicities related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500 K/cumm without granulocyte colony-stimulating factor support
  * White blood cell count ≥ 2,500 K/cumm
  * Platelets ≥ 100,000 K/cumm without transfusion
  * Hemoglobin ≥ 9.0 g/DL
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease ≤ 3.0 x IULN)
  * AST(SGOT), ALT(SGPT), and alkaline phosphatase (ALP) ≤ 3.0 x IULN; ALP ≤ 5.0 x IULN with documented bone metastases
  * Serum creatinine ≤ 2.0 x IULN or calculated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
  * Serum albumin ≥ 2.8 g/dL
  * Urine protein/creatinine ration (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)), or 24h urine protein ≤1g
  * PT/INR or PTT < 1.3 x IULN
* Castrate testosterone levels with serum testosterone ≤ 50 ng/mL at time of study drug start, with ongoing ADT throughout the study unless prior bilateral orchiectomy.
* Corrected QT interval calculated by the Fridericia formula (QTcF) ≤ 500 ms (by ECG)
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of the legally authorized representative, if applicable).
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.

Exclusion Criteria:

* Any evidence of neuroendocrine/small cell prostate cancer, or castrate resistant prostate cancer, as defined by defined by disease progression despite androgen depletion therapy (ADT), either by continuous rise in serum PSA levels as measured over at least 2 consecutive values, or the clinical or radiographic progression of disease, as assessed by the investigator.
* Prior exposure to second-generation androgen receptor inhibitors (e.g., enzalutamide, apalutamide, darolutamide).
* Prior exposure to CYP17 inhibitors (e.g. abiraterone)
* No chronic concomitant treatment with strong cytochrome P450 (CYP) 3A4 inducers or inhibitors. If patients are on such agents and these can be safely discontinued, may not have received a strong CYP3A4 inducer/inhibitor within 5 half-lives.
* Prior systemic chemotherapy for prostate cancer (either for localized or metastatic disease). Patients may have received androgen deprivation therapy (ADT) for < 12 weeks prior to start of study drug; no other cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Prior treatment with checkpoint inhibitor or other immunotherapy (e.g., anti-PD-1, anti-PD-L1, anti-CTLA4).
* Prior treatment with cabozantinib.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Inability to swallow pills.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohns disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Presence of a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 calendar days of start of study treatment. Inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Currently receiving any other investigational agents.
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardioprotection (per applicable local guidelines) and low-dose low molecular weight heparins (LMWH)
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least one week before the first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Patients with known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, nivolumab, or abiraterone or other agents used in the study.
* Uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within six months before the first dose of study treatment.

      * Subjects with a diagnosis of incidental, subsegmental PE or DVT within six months are allowed if stable, asymptomatic, and treated with anticoagulation for at least 1 week before the first dose of study treatment.
  * Gastrointestinal (GI) disorders, including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within six months before the first dose.

Note: Complete healing of an intra-abdominal abscess must be confirmed before the first dose.

* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before the first dose.
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels.
* Other clinically significant disorders that would preclude safe study participation.

  * Serious non-healing wound/ulcer/bone fracture.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).

    * Active hepatitis B or C; active HIV. Patients with well-controlled HIV or hepatitis B or C, or who have had curative treatment for hepatitis C, may be considered if they meet all other criteria and after discussion with the PI and drug manufacturers (BMS and Exelixis) using the following criteria for guidance: https://www.fda.gov/media/121319/download
    * History of organ allograft.
    * Major surgery (e.g., laparoscopic nephrectomy, GI surgery removal or biopsy of brain metastasis) within 2 weeks before the first dose of study treatment. Minor surgeries within 10 days before dose of study treatment (with the exception of the baseline biopsy, which must have occurred no less than 6 days prior to the first dose). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Patients with clinically relevant ongoing complications from prior surgery are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLTs) | Completion of 1st cycle of treatment for patients in dose level 1 & dose level 2 (estimated to be 11 months)
  * Protocol defined hematologic DLTs that occur during the first cycle that are attributed as possibly, probably, or definitely related to study treatment
  * Protocol defined non-hematologic DLTs possibly, probably, or definitely related grade 3 or 4 non-hematologic toxicity that occurs during the first cycle of treatment.

SECONDARY OUTCOMES:
PSA response rate | Through end of treatment (estimated to be 24 months)
  -Defined by at least 50% decline in PSA level from baseline measured twice at least 3 weeks apart
Overall response rate (ORR) | Through end of treatment (estimated to be 24 months)
  -Defined by proportion of patients achieving complete or partial response by RECIST 1.1 or by PCWG3 criteria
Overall survival (OS) | From start of treatment through 1 year of follow-up (estimated to be 36 months)
  -Defined as from start of treatment to date of death (all cause) or last follow-up.
Progression-free survival (PFS) | From start of treatment through 1 year of follow-up (estimated to be 36 months)
  -Defined from start of treatment to date of progression or death or last follow-up, whichever is earlier.
Disease specific survival (DSS) | From start of treatment through 1 year of follow-up (estimated to be 36 months)
  -Defined as from start of treatment to to date of death due to disease or last follow-up.
Incidence of adverse events as measured per CTCAE v 5.0 | From time of consent through 100 days after last dose of nivolumab (estimated to be 28 months)
Disease free survival (DFS) | From start of treatment through 1 year of follow-up (estimated to be 36 months)
  -Defined as from date of first PSA response or radiographic complete response to date of recurrence of disease
Duration of response (DoR) | From start of first response through 1 year of follow-up (estimated to be 36 months)
  -Defined from date of first PSA response to date of PSA progression or date of RECIST response to date of radiographic progression.

CONTACTS AND LOCATIONS:
Overall Officials: Russell K Pachynski, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu